CLINICAL TRIAL: NCT05843240
Title: Effects of Repetitive Transcranial Magnetic Stimulation on Cerebral Autoregulation in Patients With Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Vice President of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMSCA-AIS
Record Dates: First submitted 2023-04-20; First posted 2023-05-06 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Transcranial Magnetic Stimulation
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rTMS (Active Comparator): Patients are treated with repetitive transcranial magnetic stimulation (rTMS).
  Interventions: Procedure: Repetitive transcranial magnetic stimulation
- sham-rTMS (Placebo Comparator): Patients are treated with sham repetitive transcranial magnetic stimulation (sham-rTMS).
  Interventions: Procedure: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Procedure: Repetitive transcranial magnetic stimulation — After enrollment, patients received rTMS once a day for 5 consecutive days (stimulation plan: stimulation of M1 region on the affected side at 10Hz).
  Arms: rTMS
Procedure: Sham repetitive transcranial magnetic stimulation — After enrollment, patients received sham-rTMS once a day for 5 consecutive days with the same parameters as the rTMS group, but the coil was rotated 90° away from the scalp.
  Arms: sham-rTMS

SUMMARY:
The purpose of this study was to investigate the effect of repetitive transcranial magnetic stimulation on cerebral autoregulation in patients with acute ischemic stroke.

DETAILED DESCRIPTION:
Current studies have shown that repetitive transcranial magnetic stimulation can change the excitability of nerve cells, improve intracerebral artery blood supply, and even reduce the degree of neurological impairment in patients with ischemic stroke. The purpose of this study was to investigate the effect of repetitive transcranial magnetic stimulation on cerebral autoregulation in patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, both sexes;
2. Clinically definite diagnosis of acute ischemic stroke;
3. Baseline National Institute of Health Stroke Scale (NIHSS) score ≤25;
4. Pre-onset modified Rankin Scale (mRS) score ≤1;
5. Randomized and initiated transcranial magnetic stimulation within 1 week of onset;
6. Subject or legal representative agreed to the treatment and signed the informed consent.

Exclusion Criteria:

1. Presence of a medical condition such as severe cognitive impairment or mental impairment;
2. Patients with serious physical diseases or who have had craniocerebral surgery;
3. Previous history of epilepsy, family history of epilepsy or presence of seizure provoking factors;
4. Pregnancy or breastfeeding;
5. The presence of metal foreign bodies near the stimulation site, such as intracranial metal implants, cochlear implants, built-in pulse generators (brain pacemakers, cardiac pacemakers), etc.;
6. Patients who are unable to complete cerebral autoregulation, or bilateral temporal window penetration poorly;
7. life expectancy of ≤3 months or inability to complete the study for other reasons;
8. unwillingness to be followed up or poor treatment compliance;
9. Those who are participating in other clinical investigators, or who have participated in other clinical studies within 3 months prior to enrollment, or who have participated in this study;
10. Other conditions that the investigators deemed unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2023-05-07 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
phase difference(PD) in degree | 0-5 days
  A cerebral autoregulation parameter derived from transfer function analysis. Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the cerebral autoregulatory parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China